CLINICAL TRIAL: NCT06671535
Title: Effect of Kidney Replacement Therapy with Polymethylmethacrylate Membranes on Pruritus-related Quality of Life in Patients Receiving Maintenance Haemodialysis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saint Petersburg State University, Russia (Other)
Responsible Party: Principal Investigator, Ekaterina Parshina, Chief of Nephrology and Dialysis department, Saint Petersburg State University, Russia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PMMA and pruritis
Record Dates: First submitted 2024-10-31; First posted 2024-11-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-03

CONDITIONS: CKD (Chronic Kidney Disease) Stage 5D; Hemodialysis; Pruritis
Keywords: polymethylmethacrylate membranes; CKD-associated pruritis; PMMA membranes
MeSH Terms: conditions — Renal Insufficiency, Chronic; Pruritus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PMMA arm (Experimental): Patients in the experimental group will receive maintenance hemodialysis using polymetilmethacrylate membranes for 2 months.
  Interventions: Device: Polymethylmethacrylate membrane
- Polysulfone arm (Active Comparator): Patients in the control group will receive maintenance hemodialysis using polysulfone membranes for 2 months.
  Interventions: Device: polysulfone membranes

INTERVENTIONS:
Device: Polymethylmethacrylate membrane — A polymethylmethacrylate hollow fiber membrane (PMMA membrane) has unique properties including the uniform structure and the adsorption property.
  Arms: PMMA arm
Device: polysulfone membranes — Dialyzers containing polysulfone membranes are widely used for modern dialysis therapies as they allow efficient removal of a broad spectrum of uremic toxins.
  Arms: Polysulfone arm

SUMMARY:
This randomized controlled trial aims to evaluate the effect of polymethylmethacrylate dialysis membranes use on the intensity of pruritus in patients with CKD stage 5D receiving maintenance hemodialysis.

The main question it aims to answer is: Does the use of polymethylmethacrylate (PMMA) membranes reduce the intensity of pruritus in dialysis patients?

Researchers will compare PMMA membranes to standard polysulfone-based membranes to see if PMMA works to reduce moderate-to-severe pruritis and pruritis-related quality of life.

Participants will:

* receive maintenance hemodialysis with PMMA or polysulfone membranes for 2 months;
* fill in questionnaires about intensity of pruritis and its impact on daily life.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CKD stage 5D, maintenance hemodialysis not less than 3 months prior screening;
* Moderate-to-severe pruritis (WI-NRS score ≥ 4);
* Adequate dialysis dose (spKt/V≥1,4 and/or eKt/V≥1,2);
* Dialysis treatment regimen: three sessions per week of at least 4 hours duration;
* Signed informed consent.

Exclusion Criteria:

* Presence of active skin disease, cholestasis, severe secondary hyperparathyroidism and other conditions that, in the investigator's opinion, may be responsible for pruritus.
* Noncompliance of the patient with the protocol (in the investigator's opinion).
* Use of haemodiafiltration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2025-01-27 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
5D Elman Itch Scale total score | From enrollment to the end of treatment at 8 weeks
  The 5-D itch scale is a reliable, multidimensional measure of itching that has been validated in patients with chronic pruritus to able to detect changes over time. This questionnaire was designed to be useful as an outcome measure in clinical trials. The five dimensions are degree, duration, direction, disability and distribution.

SECONDARY OUTCOMES:
WI-NRS score | From enrollment to the end of treatment at 8 weeks
  24-hour Worst Itching Intensity Numerical Rating Scale
Skindex-16 score | From enrollment to the end of treatment at 8 weeks
  Multidimensional tool to assess pruritis
Itch-MOS score | From enrollment to the end of treatment at 8 weeks
  Itch-MOS questionnaire aims to evaluate impact of pruritis on sleep.
5D Elman Itch Scale total score | From the end of active treatment to the end of follow-up (4 weeks)
WI-NRS score | From the end of active treatment to the end of follow-up (4 weeks)
Skindex-16 score | From the end of active treatment to the end of follow-up (4 weeks)
Itch-MOS score | From the end of active treatment to the end of follow-up (4 weeks)
C-reactive protein concentration | From enrollment to the end of treatment at 8 weeks
Serum ferritin | From enrollment to the end of treatment at 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Petersburg State University Hospital, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: No